CLINICAL TRIAL: NCT06395207
Title: A Short Period of Proactive Community Case Management (ProCCM) to Improve Early Care-seeking for Fever in Sierra Leone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Tulane University (Other); Sustainable Health Systems Sierra Leone (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ProCCM V1 2024
Record Dates: First submitted 2024-04-23; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Health Services Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimized standard of care for CCM plus ProCCM (Experimental): ProCCM will be implemented for two months near the start of the transmission season, and the existing program will be supplemented to ensure that HTR CHWs have all commodities needed for malaria testing and treatment and are adequately trained on SBCC messages to ensure activities are implemented as designed.
  Interventions: Behavioral: Proactive community case management
- Standard of care (Active Comparator): As in arm 1 without ProCCM
  Interventions: Behavioral: Strengthened SBCC and stock out mitigation
- Routine implementation (control) (No Intervention): No changes (business as usual) to iCCM, SBCC and stock management.

INTERVENTIONS:
Behavioral: Proactive community case management — Community health workers conduct proactive visits to households in their community every two weeks for two months to screen for fever and test and treat febrile individuals for malaria.
  Arms: Optimized standard of care for CCM plus ProCCM
Behavioral: Strengthened SBCC and stock out mitigation — Ensure CHWs have all commodities needed for malaria testing and treatment and are adequately trained on SBCC messages to ensure activities are implemented as designed in the national strategy.
  Arms: Standard of care

SUMMARY:
This is a three arm cluster randomized control trial to determine if proactive community case management (ProCCM) conducted over a short period of time improves care-seeking indicators for febrile illnesses in children in hard to reach (HTR) areas of Sierra Leone compared to integrated community case management (iCCM). The three arms include:

1. Optimized standard of care for CCM plus ProCCM - ProCCM will be implemented for two months near the start of the transmission season, and the existing program will be supplemented to ensure that HTR CHWs have all commodities needed for malaria testing and treatment and are adequately trained on SBCC messages to ensure activities are implemented as designed.
2. Optimized standard of care- as in arm 1 without ProCCM
3. Routine implementation (control) - no changes (business as usual) to iCCM, SBCC and stock management.

ELIGIBILITY:
Inclusion Criteria:

* Household lives within the study cluster
* Head of household or a household member over the age of 18 provides verbal consent for the HTR CHW visit
* All available household members at the time of the HTR CHW visits are eligible to receive services

Exclusion Criteria:

* Household does not live within the study cluster
* Household does not provide consent for the study visit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of children under five years of age with recent fever (within the past two weeks) who sought care from a CHW or public health facility on the same day or day after fever onset | Cross sectional collected immediately post-intervention and 5 months post-intervention
  Changes in care seeking will be assessed through three cross-sectional surveys. A baseline survey will be conducted prior to intervention implementation followed by a second survey at or near the end of the ProCCM intervention period and a final survey at the end of the malaria transmission season.

SECONDARY OUTCOMES:
Cost per additional fever case promptly seeking care at qualified provider | 5 months post-intervention
  Using project records and information from the cross-sectional surveys, the cost of delivering ProCCM, incremental SBCC and stockout management interventions will be determined with the incremental number of fever cases receiving prompt management by a qualified provider as the denominator.
Barriers and enablers of care-seeking behavior for febrile illness of people of all ages and how ProCCM impacts this behavior explored through focus groups | End of the malaria transmission season which will be 2 months post intervention
  Focus group discussions will be held with community members post-intervention to assess barriers and enablers of care-seeking for febrile illness among people of all ages and how ProCCM impacts this behavior as reported by community members
Perceptions of the availability, cost, quality, and ease of seeking care for febrile illness explored through focus groups and in-depth interviews with community members. | End of the malaria transmission season which will be 2 months post intervention
  Focus group discussions and in-depth interviews will be held with community members to explore their perception of the intervention and how it impacts their sense of the availability, cost, quality, and ease of seeking care for febrile illness.
Job satisfaction and perceived workload as described by CHWs during focus groups and interviews | End of the malaria transmission season which will be 2 months post intervention
  Focus groups and in-depth interviews will be conducted with community health workers to explore their job satisfaction and perceived workload as it relates to the intervention.
Differences in touchpoints and connection between CHWs and health facility staff as described through qualitative analysis. | End of the malaria transmission season which will be 2 months post intervention
  In-depth interviews will be conducted with health facility staff and peer supervisors to explore how the intervention influences their perceived linkages and touchpoints with CHWs.

IPD SHARING:
Plan to Share IPD: No